CLINICAL TRIAL: NCT01042912
Title: A Single-centered Investigation Into the Frequency Domain Patterns in the Carotid Vessel in Patients With Suspected Stenosis
Brief Title: Frequency Analysis of Carotid Artery Disease
Status: Withdrawn | Type: Observational
Why Stopped: PI left inistitution
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 901M57884
Record Dates: First submitted 2010-01-04; First posted 2010-01-06 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Carotid Artery Disease
Keywords: diagnosis; carotid; artery; disease; auscultation; sound
MeSH Terms: conditions — Carotid Artery Diseases; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine if carotid artery stenosis can be detected using an electronic stethoscope. This study will use a commercially available electronic stethoscope to record carotid sounds in patients with suspected carotid artery stenosis. The presence of absence of abnormal vessels will be confirmed by diagnostic ultrasound as part of normal patient care at this institution.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-80
* Indicated for diagnostic ultrasound related to carotid artery stenosis

Exclusion Criteria:

* Pregnant women
* Prior carotid intervention

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any inpatient or outpatient with inclusion criteria met and exclusion criteria not met presenting for aniography to the University of Minnesota Fairview Hospital or Clinic in Minneapolis or Redwing, Minnesota
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-05; Primary Completion 2010-02 (Estimated); Study Completion 2010-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Marie A Johnson, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical Center (UMMC) Fairview Clinics, Minneapolis, Minnesota, United States